CLINICAL TRIAL: NCT04751084
Title: Use of Buscopan in Patients Undergoing IVF/Intracytoplasmic Sperm Injection Treatment With High and Low Uterine Contraction Frequency Prior to Embryo Transfer: A Prospective Double-blinded Randomized Controlled Trial
Brief Title: Buscopan in Patients Undergoing IVF/Intracytoplasmic Sperm Injection Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Mak Sze Man Jennifer, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019.109-T
Record Dates: First submitted 2021-01-26; First posted 2021-02-11 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: IVF; Intracytoplasmic Sperm Injection
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: A prospective double blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blinded to the randomization list
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Active Comparator): 20mg Buscopan intravenous will be given 5 minutes prior to embryo transfer
  Interventions: Drug: Buscopan 20 milligrams/ML Injectable Solution
- control group (Placebo Comparator): 2ml Normal Saline intravenous will be given 5 minutes prior to embryo transfer
  Interventions: Drug: Buscopan 20 milligrams/ML Injectable Solution

INTERVENTIONS:
Drug: Buscopan 20 milligrams/ML Injectable Solution — cases will be randomized to Buscopan group or Normal Saline group, injection will be given 5 minutes prior to embryo transfer
  Other Names: Normal Saline

SUMMARY:
To determine if the use of Buscopan in patients undergoing IVF/ICSI treatment with high uterine contraction frequency prior to embryo transfer has a higher live birth rate.

ELIGIBILITY:
Inclusion Criteria:

- Women undergoing embryo transfer in either fresh or frozen cycles

Exclusion Criteria:

* Women aged > 42 years old
* Women with factors which will affect uterine contractility
* congenital uterine anomaly
* acquired uterine pathology such as myoma >5cm, adenomyosis >5cm or endometrial polyp
* Women with presence of hydrosalpinx
* Women undergoing pre-implantation genetic test in IVF cycles
* History of allergy to misoprostol , Buscopan® or same group of drug
* Contraindication to the use of Buscopan® e.g. glaucoma, myasthenia gravis, tachycardia, megacolon
* Women who are on other smooth muscle relaxant other than Buscopan®

Max Age: 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — aged <42 years old
Enrollment: 675 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-09-14 (Estimated)

PRIMARY OUTCOMES:
live birth rate | after 24 weeks of gestation
  live baby born

SECONDARY OUTCOMES:
implantation rate | 8-10 days after embryo transfer
  positive pregnancy test
clinical pregnancy rate | at 6 weeks gestation
  the presence of at least one gestational sac
multiple pregnancy rate | after 24 weeks of gestation
  more than 1 live birth
miscarriage rate | before 24 weeks of gestation
  biochemical if there is no US evidence of pregnancy and clinical if there is US evidence of pregnancy
ectopic pregnancy rate | at 6-7 weeks of gestation
  IU sac out of uterine cavity

CONTACTS AND LOCATIONS:
Overall Officials: SZE MAN JENNIFER MAK, Principal Investigator — Chinese University of Hong Kong; NGA PING PATRICIA IP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong